CLINICAL TRIAL: NCT00309062
Title: A Multicentre Randomised Placebo-controlled Double-blind Clinical Trial for Evaluation of Safety and Efficacy of Immunotherapy With an Aluminium Hydroxide-adsorbed Recombinant Hypoallergenic Derivative of the Major Birch Pollen Allergen, Bet v 1
Brief Title: Safety and Efficacy of Recombinant Birch Pollen Allergen in the Treatment of Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Al0103rB
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Birch Pollen Allergy
Keywords: Allergy; Birch pollen; Recombinant
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Recombinant birch pollen

SUMMARY:
Safety and efficacy of recombinant birch pollen allergen in the treatment of allergic rhinoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Positive Skin Prick Test reaction to birch pollen
* Positive RAST result to birch pollen
* Positive Provocation Test result to birch pollen

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-12; Primary Completion 2006-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M D, Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de